CLINICAL TRIAL: NCT04161144
Title: Enhancing Self-regulation by Altering Memories That Increase Risk of Relapse Among Smokers: A Translational Clinical Neuroscience Study of a Novel Medication
Brief Title: Enhancing Self Regulation Among Smokers
Acronym: MIMIC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 76669
Record Dates: First submitted 2019-11-08; First posted 2019-11-13 (Actual); Results first posted 2021-03-09 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Smoking Cessation; Smoking, Cigarette; Nicotine Dependence
MeSH Terms: conditions — Smoking Cessation; Cigarette Smoking; Tobacco Use Disorder | interventions — Sirolimus; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rapamycin 15mg (sirolimus) (Active Comparator): Participants will receive three 5mg pills from a nurse in the Research Nexus, some participants will receive the study medication and others will be randomized to the placebo control group.
  Interventions: Drug: sirolimus
- Placebo (Placebo Comparator): Participants will receive three 5mg pills from a nurse in the Research Nexus, some participants will receive the study medication and others will be randomized to the placebo control group.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: sirolimus — Rapamycin (sirolimus) is administered in three 5mg oral capsules. This administration happens once during the first visit.
  Other Names: rapamycin; rapamune
  Arms: Rapamycin 15mg (sirolimus)
Drug: Placebo — Placebo is administered in three 5mg oral capsules. This administration happens once during the first visit.
  Other Names: Sugar Pill
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the effects of rapamycin (sirolimus) versus a placebo, an inactive substance, on responses to smoking cues in individuals with nicotine dependence. Rapamycin (sirolimus) is a FDA-approved antibiotic and immunosuppressive drug that is currently used to (a) prevent organ transplant recipients from rejecting their transplants (b) treat cardiovascular diseases, and (c) treat some forms of cancer. Rapamycin (sirolimus) is not FDA-approved for smoking cessation. The use of rapamycin (sirolimus) in this study is investigational, meaning that the study medication is not a proven treatment for nicotine dependence, however this study will examine the medication's use as a potential future treatment for nicotine dependence.

DETAILED DESCRIPTION:
The proposed study will employ 58 ND treatment-seeking smokers who will be randomly assigned to receive either 15-mg of sirolimus or placebo (group n's=29) immediately after the first of two smoking cue exposure sessions scheduled to occur on consecutive days. The first session will serve as a Retrieval session during which smoking (e.g., handling and lighting of a cigarette) cue exposure will elicit retrieval and reconsolidation of smoking-related memories; the second session will be a Test session to examine the potential modulatory role of sirolimus on the reconsolidation of memories putatively elicited during the retrieval session. Participants will be required to refrain from smoking the night before (bedtime) their first laboratory (i.e., Retrieval) session and will remain abstinent from smoking until the completion of the second laboratory (i.e., Test) session. It is posited that changes in reactivity during the test session will reflect medication effects on memory reconsolidation that occurred following the retrieval session. Measures of subjective responses (i.e., craving) and physiological reactivity (i.e., heart rate & skin conductance) will be obtained before, during and after cue presentations in both sessions. The durability of any observed treatment effects will be assessed in a Follow-up session performed 7-days following completion of the test session. Treatment effects on self-report measures of smoking behavior during the 7-days preceding the Follow-up session will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Participants must smoke 10+ cigarettes/day for three or more years
* Have a Fagerström Test for Nicotine Dependence score greater than or equal to 4
* Be willing to make a cessation attempt
* Willing to comply with reinforced abstinence requirements for the three laboratory sessions
* Willing to use appropriate birth control methods during study participation including oral contraceptives, barrier methods (diaphragm or condoms with spermicide or both), surgical sterilization, use of an intra-uterine contraceptive device, or complete abstinence from sexual intercourse
* Remain abstinent from alcohol and all non-prescription drugs prior to medication administration and testing sessions
* Live with within a 50 mile radius of our research program and have reliable transportation
* Consent to fast for a two-hour period prior to medication administration
* Consent to random assignment to rapamycin (sirolimus) vs. placebo conditions

Exclusion Criteria:

* Dependence on other substances (may meet criteria for abuse)
* Undergoing other smoking cessation treatment (e.g., nicotine replacement, Chantix)
* Taking medications that may interact with the study medication or alter responding on any study measure
* Are pregnant, nursing, or of childbearing potential and not using birth control
* Present evidence of or a history of significant endocrine, cardiovascular, pulmonary, renal or neurological disease, as these conditions may affect heart rate or skin conductance measurement
* Have significant liver impairment (as indicated by alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) values that are three times the upper limit of normal) as rapamycin (sirolimus) is hepatically metabolized
* Have an existing infection or immune system disorder as rapamycin (sirolimus) has known immunosuppressive properties
* Have a history of or current psychotic disorder, severe major depression as evidenced by active and profound psychomotor retardation and/or persistent and intense suicidal ideation
* Currently taking anti-arrhythmic agents, psychostimulants or any other agents known to interfere with heart rate and skin conductance monitoring
* Have known or suspected hypersensitivity to macrolide compounds (such as rapamycin/sirolimus)
* Taking medications that could adversely interact with study medication including but not limited to significant inhibitors of CYP2D6 or CYP3A4 (voriconazole, fluconazole, itraconazole, erythromycin, clarithromycin, diltiazem, verapamil, etc.) or significant inducers of CYP3A4, such as anticonvulsants (carbamazepine, phenobarbital, phenytoin, etc.) and antibiotics (rifabutin, rifapentine, etc.)
* Have a history of thrombocytopenia, idiopathic thrombocytopenia purpura (ITP), or with a current platelet count of less than 100,000 cells per mm3,
* Have any unhealed wounds, including but not limited to oral ulcers, foot ulcers, or recent surgical or trauma wounds
* Have any planned surgeries within the next month, including surgical dental procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Saladin, Ph.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rapamycin 15mg (Sirolimus) | Placebo
Started | 12 | 10
Completed | 11 | 9
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rapamycin 15mg (Sirolimus) | Placebo | Total
Number analyzed (Participants) | 12 | 10 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (11.3) | 47.1 (15.2) | 49.4 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 9 | 8 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 1 | 5
  White | 8 | 8 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 10 | 22
Cigarettes Per Day [Mean (Standard Deviation); unit: Cigarettes Per Day] — Cigarettes per day noted as 90-day average as reported on the Time-Line-Follow-Back. 90 days prior to study baseline.
  Cigarettes Per Day | 21.5 (9.5) | 19.7 (10.3) | 20.7 (9.7)

OUTCOME MEASURES:

1. Primary Outcome: Craving Levels in Response to Cue
Description: Patients are asked about craving level on a scale of 0-100, 0 is least amount of craving and 100 is highest amount of craving
Time Frame: Study visit 1 (Baseline; day 0), visit 2 (day 7) and visit 3 (day 14)
Population: Data entered are the number of participants under the cue condition at study visit 1 (Baseline; day 0), visit 2 (day 7) and visit 3 (day 14)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rapamycin 15mg (Sirolimus) | Placebo
Number analyzed (Participants) | 12 | 9
score on a scale
  Day 0: Pre-Cue | 69.6 (26.3) | 66.3 (27.8)
  Day 0: Cue | 56.1 (35.2) | 74.4 (16.1)
  Day 0: Cue+0 min | 62.6 (34.4) | 83.2 (18.1)
  Day 0: Cue+10 min | 53.1 (33.4) | 72.8 (16.8)
  Day 0: Cue+20 min | 50.4 (37.7) | 71.7 (23.5)
  Day 0: Cue+30 min | 44.3 (37.7) | 67.8 (25.9)
  Day 0: Cue+40 min | 39.1 (39.7) | 67.2 (27.6)
  Day 0: Cue+50 min | 38.1 (37.7) | 63.7 (32.1)
  Day 7: Pre-Cue: number analyzed (Participants) | 11 | 9
  Day 7: Pre-Cue | 40.9 (37.6) | 62.2 (27.7)
  Day 7: Cue: number analyzed (Participants) | 11 | 9
  Day 7: Cue | 41.9 (38.1) | 67.2 (29.3)
  Day 7: Cue+0 min: number analyzed (Participants) | 11 | 9
  Day 7: Cue+0 min | 46.8 (36.1) | 68.3 (28.7)
  Day 7: Cue+10 min: number analyzed (Participants) | 11 | 9
  Day 7: Cue+10 min | 43.1 (37.2) | 59.4 (27.4)
  Day 7: Cue+20 min: number analyzed (Participants) | 11 | 9
  Day 7: Cue+20 min | 43.4 (37.9) | 55.5 (29.6)
  Day 7: Cue+30 min: number analyzed (Participants) | 11 | 9
  Day 7: Cue+30 min | 40.4 (40.0) | 52.8 (30.7)
  Day 7: Cue+40 min: number analyzed (Participants) | 11 | 9
  Day 7: Cue+40 min | 39.8 (40.5) | 52.2 (31.0)
  Day 7: Cue+50 min: number analyzed (Participants) | 11 | 9
  Day 7: Cue+50 min | 39.7 (40.6) | 49.4 (33.2)
  Day 14: Pre-Cue: number analyzed (Participants) | 11 | 9
  Day 14: Pre-Cue | 37.3 (36.8) | 41.7 (31.1)
  Day 14: Cue: number analyzed (Participants) | 11 | 9
  Day 14: Cue | 45 (34.5) | 46.7 (32.3)
  Day 14: Cue+0 min: number analyzed (Participants) | 11 | 9
  Day 14: Cue+0 min | 44.3 (34.5) | 48.9 (32.1)
  Day 14: Cue+10 min: number analyzed (Participants) | 11 | 9
  Day 14: Cue+10 min | 43.6 (32.4) | 45.6 (29.5)
  Visit 3: Cue+20 min: number analyzed (Participants) | 11 | 9
  Visit 3: Cue+20 min | 40.3 (32.1) | 40 (28.6)
  Day 14: Cue+30 min: number analyzed (Participants) | 11 | 9
  Day 14: Cue+30 min | 39.5 (32.7) | 43.3 (31.2)
  Day 14: Cue+40 min: number analyzed (Participants) | 11 | 9
  Day 14: Cue+40 min | 40.5 (32.3) | 38.9 (30.7)
  Day 14: Cue+50 min: number analyzed (Participants) | 11 | 9
  Day 14: Cue+50 min | 41.2 (33.1) | 37.2 (30.1)

2. Primary Outcome: Heart Rate in Response to Cue
Description: Heart rate is measured using a Biopac machine and Acqknowledge software at different timepoints throughout each visit while the participants are exposed to smoking cues.
Time Frame: Study visit 1 (Baseline; day 0), visit 2 (day 7) and visit 3 (day 14)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Rapamycin 15mg (Sirolimus) | Placebo
Number analyzed (Participants) | 12 | 10
Beats per minute
  Day 0: Pre-Cue: number analyzed (Participants) | 12 | 9
  Day 0: Pre-Cue | 72 (9) | 75 (16)
  Day 0: Cue+0 min: number analyzed (Participants) | 12 | 9
  Day 0: Cue+0 min | 71 (11) | 73 (13)
  Day 0: Cue+10 min: number analyzed (Participants) | 12 | 9
  Day 0: Cue+10 min | 69 (12) | 70 (14)
  Day 0: Cue+20 min: number analyzed (Participants) | 12 | 9
  Day 0: Cue+20 min | 69 (11) | 69 (15)
  Day 0: Cue+30 min: number analyzed (Participants) | 12 | 9
  Day 0: Cue+30 min | 70 (13) | 72 (12)
  Day 0: Cue+40 min: number analyzed (Participants) | 12 | 9
  Day 0: Cue+40 min | 71 (11) | 68 (12)
  Day 0: Cue+50 min: number analyzed (Participants) | 12 | 9
  Day 0: Cue+50 min | 72 (11) | 70 (11)
  Day 7: Pre-Cue: number analyzed (Participants) | 12 | 9
  Day 7: Pre-Cue | 73 (9) | 75 (11)
  Day 7: Cue+0 min: number analyzed (Participants) | 12 | 9
  Day 7: Cue+0 min | 71 (11) | 74 (11)
  Day 7: Cue+10 min: number analyzed (Participants) | 12 | 9
  Day 7: Cue+10 min | 69 (11) | 75 (9)
  Day 7: Cue+20 min: number analyzed (Participants) | 12 | 9
  Day 7: Cue+20 min | 71 (10) | 74 (12)
  Day 7: Cue+30 min: number analyzed (Participants) | 12 | 9
  Day 7: Cue+30 min | 71 (12) | 74 (14)
  Day 7: Cue+40 min: number analyzed (Participants) | 12 | 9
  Day 7: Cue+40 min | 71 (13) | 71 (12)
  Day 7: Cue+50 min: number analyzed (Participants) | 12 | 9
  Day 7: Cue+50 min | 70 (12) | 72 (14)
  Day 14: Pre-Cue: number analyzed (Participants) | 11 | 10
  Day 14: Pre-Cue | 75 (7) | 73 (14)
  Day 14: Cue+0 min: number analyzed (Participants) | 11 | 10
  Day 14: Cue+0 min | 70 (15) | 73 (17)
  Day 14: Cue+10 min: number analyzed (Participants) | 11 | 10
  Day 14: Cue+10 min | 70 (15) | 66 (14)
  Day 14: Cue+20 min: number analyzed (Participants) | 11 | 10
  Day 14: Cue+20 min | 71 (11) | 66 (14)
  Day 14: Cue+30 min: number analyzed (Participants) | 11 | 10
  Day 14: Cue+30 min | 73 (9) | 68 (15)
  Day 14: Cue+40 min: number analyzed (Participants) | 11 | 10
  Day 14: Cue+40 min | 72 (13) | 68 (16)
  Day 14: Cue+50 min: number analyzed (Participants) | 11 | 10
  Day 14: Cue+50 min | 72 (10) | 70 (16)

3. Secondary Outcome: Average Cigarettes Smoked Per Day
Description: Patients will be asked how many cigarettes per day they smoked 90 days prior to starting the study. Patients are then given a smoking and alcohol diary to complete during the course of the trial.
Time Frame: Visit 1 through Visit 3 (day 0-day 14)
Population: Self-reported average cigarettes smoked per day reported between study visit 1 and visit 3
Measure: Mean (Standard Deviation); unit: Cigarettes Per Day
Arm/Group | Rapamycin 15mg (Sirolimus) | Placebo
Number analyzed (Participants) | 11 | 9
Cigarettes Per Day | 7.6 (6.2) | 13.5 (9.5)

ADVERSE EVENTS:
Time Frame: 14 days
Arm/Group | Rapamycin 15mg (Sirolimus) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/10
Other Adverse Events (participants affected / at risk) | 6/12 | 5/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rapamycin 15mg (Sirolimus) (N=12) | Placebo (N=10)
Headache (Nervous system disorders) | 5 (8) | 2 (2)
Dry Mouth (General disorders) | 1 (3) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Taste Anomoly (General disorders) | 1 (2) | 1 (2)
Increased Thirst (General disorders) | 2 (3) | 2 (2)
Restlessness (Psychiatric disorders) | 2 (2) | 1 (1)
weakness/Fatigue (General disorders) | 2 (2) | 0 (0)
Nightmares/Vivid Dreams (Psychiatric disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-29): https://cdn.clinicaltrials.gov/large-docs/44/NCT04161144/Prot_SAP_000.pdf